CLINICAL TRIAL: NCT00261027
Title: A Pilot, Phase II, Single Center, Non-comparative, Open-label Study of Aromasin (Exemestane) in Patients With Recurrent or Refractory Stage II - IV Epithelial Ovarian Cancer
Brief Title: Aromasin (Exemestane) in Patients With Recurrent or Refractory Stage II - IV Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Dr Shailendra Verma, Ottawa Hospital Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002521-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Exemestane

SUMMARY:
This project is a pilot, phase II, open-label, single-center, non-comparative clinical study evaluating the antitumor efficacy and tolerability of exemestane in treating adult post-menopausal women with recurrent or refractory, stage II-IV, epithelial ovarian cancer.

To evaluate the efficacy and tolerability of exemestane in this population, patients will be enrolled at a single site, namely the Ottawa Regional Cancer Center. Patients selected according to the criteria outlined will receive exemestane (25 mg/day given orally once daily) until disease progression or until study withdrawal. These patients will be treated on an out-patient basis. There is no specific wash-out time required for patients who have previously received either cis or carboplatinum; however, this previous therapy must stop upon patient inclusion into this trial.

In 1st stage if less than 2/15 patients achieve a response then study will be terminated. In 2nd stage if greater than 7/28 patients achieve a response then no further investigation of the drug is warranted.Treatment (including drug dosages) A commercial supply of exemestane (Aromasin) will be provided. The medication will be administered by the patient at home (25 mg taken orally once daily until disease progression) The medication should be taken each day after a meal at the same time of the day. There are no patient diaries and no need for the patient to record the time of administration.

DETAILED DESCRIPTION:
This project is a pilot, phase II, open-label, single-center, non-comparative clinical study evaluating the antitumor efficacy and tolerability of exemestane in treating adult post-menopausal women with recurrent or refractory, stage II-IV, epithelial ovarian cancer.

To evaluate the efficacy and tolerability of exemestane in this population, patients will be enrolled at a single site, namely the Ottawa Regional Cancer Center. Patients selected according to the criteria outlined will receive exemestane (25 mg/day given orally once daily) until disease progression or until study withdrawal. These patients will be treated on an out-patient basis. There is no specific wash-out time required for patients who have previously received either cis or carboplatinum; however, this previous therapy must stop upon patient inclusion into this trial. In 1st stage if less than 2/15 patients achieve a response then study will be terminated. In 2nd stage if greater than 7/28 patients achieve a response then no further investigation of the drug is warranted.

Treatment (including drug dosages) A commercial supply of exemestane (Aromasin) will be provided. The medication will be administered by the patient at home (25 mg taken orally once daily until disease progression) The medication should be taken each day after a meal at the same time of the day. There are no patient diaries and no need for the patient to record the time of administration.

ELIGIBILITY:
Inclusion Criteria:

* · Patients aged 18 years or older with a documented diagnosis of metastatic, stage II-IV, epithelial ovarian cancer and a histological/cytological confirmation of disease.· Patients must be oophorectomized or be post-menopausal (i.e. no menses within the last 12 months).· Patients should have objective evidence of measurable disease according to the modified RECIST guidelines. If no measurable disease is present, there must be a CA 125 level of ³ 30 U/mL in combination with non-measurable disease and/or ascites.· Patients may be designated:· First line - patients who have either refused or did not qualify for initial therapy with standard cis- or carboplatin + paclitaxel.· Refractory - progression while on chemotherapy, or relapse within 12 months of final chemotherapy (with a maximum of 2 lines of chemotherapy treatment)· Recurrent - relapse beyond 12 months of final chemotherapy (with a maximum of 2 lines of chemotherapy treatment)· In patients having received radiation therapy, at least 4 weeks must have passed subsequent to the cessation of the radiation therapy, prior to the baseline assessment in this study.· Patients with ECOG performance status of 0, 1 or 2 and a life expectancy of > 3 months.· Patients must have adequate haematological (WBC ³ 4000/mL, neutrophils ³ 2000/mL, platelets ³ 100,00/mL), hepatic (total bilirubin £ 1.5 x upper limit normal (ULN), AST/ALT £ 3 x ULN)) and renal (serum creatinine < 1.5 X ULN) organ functions.· Patients must give written informed consent signed prior to registration.

Exclusion Criteria:

* Known hypersensitivity to exemestane· Participation in another clinical study within thirty days prior to the treatment on this study. Concurrent treatment with other experimental drugs or anticancer therapy.· Patients with rapidly progressive disease for which hormonal therapy may not be indicated.· Concomitant malignancies except for adequately treated carcinoma in situ of the uterine cervix or basal or squamous cell carcinoma of the skin. Patients with other malignancies must be disease free for at least 5 years.· Patients with metastatic disease of the central nervous system, eg. Paraneoplastic cerebellar degeneration, metastatic medulloblastoma, intramedullary spinal cord involvement, etc.· Patients having received prior hormonal therapy for ovarian cancer including tamoxifen and aromatase inhibitors.· Patients with any other concurrent disease, which in the opinion of the Investigator, would make the patient inappropriate for entry into this study.· Patients who are not accessible for treatment and follow-up in scheduled hours at the participating center.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-01; Primary Completion 2007-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
response rate toxicities

SECONDARY OUTCOMES:
-Time to detectable virus in the Alvac alone group and the placebo group. -Time to rebound of plasma HIV RNA level to 10,000 copies/ml -Viral set-point -Magnitude of viral rebound -HIV-specific immune function at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fung Kee Fung, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Regional Cancer Center, Ottawa, Ontario, Canada